CLINICAL TRIAL: NCT04452058
Title: CT-based Radiomic Algorithm for Assisting Surgery Decision and Predicting Immunotherapy Response of NSCLC
Acronym: TOP-RLC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Herui Yao, Principal Investigator, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SYSEC-KY-KS-2019-107
Record Dates: First submitted 2020-06-25; First posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Predictive Cancer Model; Lung Cancer; Preinvasive Adenocarcinoma
Keywords: Radiomics; Early stage; Pulmonary nodule; Pericancerous tissue; Immunotherapy
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma in Situ

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Internal cohort: The internal cohort was retrospective enrolled in Guangdong Provincial People's hospital from March 1, 2015 to December 31,2019. Patients with single pulmonary lesion underwent preoperative chest CT scan and histologically confirmed precancerous lesions or early stage lung adenocarcinoma after thoracic surgery was included.
  Interventions: Other: Radiomic Algorithm
- External cohort 1: The same inclusion/exclusion criteria were applied for another independent centers, Sun Yat-sen Memorial Hospital ,Guangdong Province, China, forming an external validation cohort of 73 patients
  Interventions: Other: Radiomic Algorithm
- External cohort 2: The same inclusion/exclusion criteria were applied for another independent centers, Zhoushan Lung Cancer Institution, Zhejiang Province, China, forming second external validation cohort of 30 patients
  Interventions: Other: Radiomic Algorithm
- Immune Cohort: The internal cohort was retrospective enrolled in Guangdong Provincial People's hospital from March 1, 2015 to May 31,2020. Patients with advanced lung cancer underwent preoperative chest CT scan and histologically confirmed NSCLC before receiving immunotherapy was included.
  Interventions: Other: Radiomic Algorithm

INTERVENTIONS:
Other: Radiomic Algorithm — Different radiomic and machine learning strategies for radiomic features extraction, sorting features and model constriction

SUMMARY:
The purpose of this study was to investigate whether the combined radiomic model based on radiomic features extracted from focus and perifocal area (5mm) can effectively improve prediction performance of distinguishing precancerous lesions from early-stage lung adenocarcinoma, which could assist clinical decision making for surgery indication. Besides, response and long term clinical benefit of immunotherapy of advanced NSCLC lung cancer patients could also be predicted by this strategy.

DETAILED DESCRIPTION:
Early detection and diagnosis of pulmonary nodules is clinically significant regarding optimal treatment selection and avoidance of unnecessary surgical procedures. Deferential pathology results causes widely different prognosis after standard surgery among pulmonary precancerous lesion, atypical adenomatous hyperplasia (AAH) as well as adenocarcinoma in situ (AIS), and early stage invasive adenocarcinoma (IAC). The micro-invasion of pulmonary perifocal interstitium is difficult to identify from AIS unless pathology immunohistochemical study was implemented after operation，which may causes prolonged procedure time and inappropriate surgical decision-making. Key feature-derived variables screened from CT scans via statistics and machine learning algorithms, could form a radiomics signature for disease diagnosis, tumor staging, therapy response adn patient prognosis. The purpose of this study was to investigate whether the combined radiomic signature based on the focal and perifocal（5mm）radiomic features can effectively improve predictive performance of distinguishing precancerous lesions from early stage lung adenocarcinoma. Besides, immunotherapy response is various among patients and no more than 20% of patients could benefit from it. None reliable biomarker has been found yet expect Programmed death-ligand 1 (PD-L1) expression, the only approved biomarker for immunotherapy. However recent reports suggested that patients could benefit from immunotherapy regardless of PD-L1 positive or negative. On the contrast, radiomics has show it advantages of non-invasiveness, easy-acquired and no limitation of sampling. Therefore, we applied this strategy in prediction for the immunotherapy response of advanced NSCLC lung cancer patients receiving immune checkpoint inhibitors (ICIs), which would prevent some non-benefit patient from the adverse effect of ICIs.

ELIGIBILITY:
Inclusion Criteria:

* (a) that were pathologically confirmed as precancerous lesions or Stage I lung adenocarcinoma （≤3cm）
* (b) standard Chest CT scans with or without contrast enhancement performed <3 months before surgery；
* (c) availability of clinical characteristics.

Exclusion Criteria:

* (a) preoperative therapy (neoadjuvant chemotherapy or radiotherapy) performed,
* (b) suffering from other tumor disease before or at the same time.
* (c) Contain other pathological components such as squamous cell lung carcinoma (SCC) or small cell lung carcinoma (SCLC) or
* (d) poor image quality.

Inclusion Criteria of immunotherapy cohort:

* (a) that were diagnosed as advanced NSCLC
* (b) Both standard Chest CT scans with contrast enhancement performed <3 months before and after first dose of immunotherapy are available；
* (c) availability of clinical characteristics.

Exclusion Criteria of immunotherapy cohort:

* (a) Ever receiving pulmonary operation on the same side of the lesion.
* (b) suffering from other tumor disease before or at the same time.
* (c) Contain other pathological components( SCLC or lymphoma) or
* (d) poor image quality.
* (e) incomplete clinical data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in Guangdong Provincial People's hospital from March 1, 2015 to May 31,2022.
  Patients from Sun Yat-sen Memorial Hospital ,Guangdong Province, China ; Zhoushan Lung Cancer Institution,Zhejiang Province,China during 2019.01-2022.3
  All Patients should be histologically confirmed NSCLC and those have preoperative chest CT scan.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Pathological subtype | 5 years
  Pathological type of pulmonary nodules
Objective Response Rate (ORR) | 5 years
  Rate of ORR in all subjects for the patients who receiving immunotherapy
Progression-free survival (PFS) | 5 years
  From enrollment to progression or death (for any reason) in immunotherapy cohort

SECONDARY OUTCOMES:
Overall survival (OS) | 5 years
  From enrollment to death (for any reason) in immunotherapy cohort
Clinical Benefit Rate (CBR) | 5 years
  Rate of CBR greater than or equal to 24 weeks in all subjects

CONTACTS AND LOCATIONS:
Overall Officials: Haiyu Zhou, PhD, Study Chair — Guangdong Provincial People's Hospital; Luyu Huang, Principal Investigator — Guangdong Provincial People's Hospital; Herui Yao, PhD, Study Director — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Yunfang Yu, Study Director — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Hanbo Cao, PhD, Study Director — Zhoushan Lung Cancer Institution
Locations (3):
- China (3):
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - Zhoushan Lung Cancer Institution, Zhoushan, Zhejiang

IPD SHARING:
Plan to Share IPD: No
The datasets used or analysed during the current study are available from the corresponding author on reasonable request.